CLINICAL TRIAL: NCT06352242
Title: La Trogocytose Est-elle un Marqueur prédictif de la réponse Aux Cellules CAR-T Dans Les Lymphomes Diffus à Grandes Cellules B ?
Brief Title: Is Trogocytosis a Predictive Marker of CAR-T Cell Response in Diffuse Large B-cell Lymphoma?
Acronym: CARTROG
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RECHMPL24_0076; 2024-A00508-39 (Registry Identifier: ID RCB)
Record Dates: First submitted 2024-03-26; First posted 2024-04-08 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-01

CONDITIONS: Diffuse Large B Cell Lymphoma
Keywords: lymphoma; chimeric antigen receptor T-cell; trogocytosis; prognosis
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patients (Other): Blood sample for Flow cytometry analysis
  Interventions: Other: Flow cytometry analysis to determine the level of trogocytosis by effector immune cells in patients
- healthy volunteer donor (Other): Blood sample for Flow cytometry analysis
  Interventions: Other: Flow cytometry analysis to determine the level of trogocytosis by effector immune cells in volunteers

INTERVENTIONS:
Other: Flow cytometry analysis to determine the level of trogocytosis by effector immune cells in patients — For each patient, a blood sample will be taken at D0 before the CAR-T cells are injected then at D3, D7, D10, D30 after the injection. Flow cytometry analysis will be performed on each sample on the day of collection to determine the level of trogocytosis by effector immune cells (T lymphocytes, NK cells, CAR-T cells) and to define the phenotypic "signature" of trogocytosis.
  Arms: Patients
Other: Flow cytometry analysis to determine the level of trogocytosis by effector immune cells in volunteers — For each healthy volunteer, a single blood sample will be taken at enrollment. Flow cytometry analysis will be performed on each sample on the day of collection to determine the level of trogocytosis of normal lymphocytes and NK cells.
  Arms: healthy volunteer donor

SUMMARY:
CAR-T cell therapy has improved survival in patients with relapsed or refractory diffuse large B-cell lymphoma (DLBCL R/R). However, only 65% of patients achieve a complete metabolic response after this treatment. To date, there is no predictive test for therapeutic response after injection of CAR-T cells. Recent studies have shown that the level of trogocytosis by immune cells correlates with the persistence of tumor cells in patients with hematological malignancies. Our main objective is to identify a phenotypic "signature" of trogocytosis predictive of therapeutic response 6 months after injection of CAR-T cells for DLBCL.

DETAILED DESCRIPTION:
The therapeutic use of CAR-T cells (Chimeric Antigen Receptor T-cells) has significantly improved the survival of patients with relapsed or refractory (R/R) diffuse large B-cell lymphoma (DLBCL). However, only 65% of patients achieve metabolic complete response after this treatment, and one year after CAR-T cells infusion, between 50 and 60% of patients have relapsed or died. Injection of CAR-T cells can also be responsible for serious immunologic and hematologic adverse events. To date, there is no predictive test for the therapeutic response or toxicity following injection of CAR-T cells.

Trogocytosis is a physiological mechanism by which an effector immune cell integrates fragments of the membrane of target cells into its membrane. These aberrant membrane markers can directly modify the functions of the cell that has acquired them. Although the physiological role of trogocytosis remains debated, recent studies have shown that the level of trogocytosis in immune effector cells is correlated with persistent tumor cells in patients with hematological malignancies.

Our main hypothesis is that, in DLBCL, the level of early trogocytosis, assessed by the aberrant expression of tumor markers on the surface of CAR-T cells and other immune effector cells between D0 and D30 after CAR-T cells infusion, correlates with therapeutic response at M6 and/or the occurrence of immunological or severe hematological CAR-T cells side-effects.

ELIGIBILITY:
Inclusion Criteria:

* For patients

  * Patient who has given free and informed consent in writing for inclusion in the non-interventional CART-BANK protocol, and orally for the CARTROG protocol,
  * Patients over 18 years of age at the time of inclusion,
  * Diagnosis of LDGCB,
  * Decision to treat with anti-CD19 CAR-T cells,
  * Patient affiliated to or benefiting from a social security scheme.
* For healthy volunteers:

  * Given free and informed oral consent for inclusion in the CARTROG protocol,
  * Donor between 18 and 70 years of age at the time of inclusion,
  * No history of solid cancer or hematological malignancy,
  * No known chronic pathology (e.g. hypertension, diabetes, etc.) and no daily treatment,
  * No surgical treatment within the last 6 months.

Exclusion Criteria:

* Patients who do not meet all the inclusion criteria,
* Pregnant or breast-feeding patient,
* Patient unable to follow the procedures and/or frequency of visits planned in the trial, for psychological, family, social or geographical reasons,
* Patient unable to consent freely to inclusion, under guardianship, curatorship or safeguard of justice.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 85 (Estimated)
Dates: Start 2024-05-22 (Actual); Primary Completion 2026-05-22 (Estimated); Study Completion 2026-05-22 (Estimated)

PRIMARY OUTCOMES:
Identification of a phenotypic "signature" of trogocytosis predictive of failure to achieve a complete metabolic response for patients with diffuse large B-cell lymphoma. | During 6 months after CAR-T cells injection
  Using flow cytometry to determine the level of trogocytosis, the phenotypic "signature" of trogocytosis will be assessed by the AUC : area under the ROC (Receiver operating characteristic) curve; established on circulating CAR-T cells, T lymphocytes and NK cells of patients, and defined as: the percentage of cells aberrantly expressing different tumor antigens normally expressed on lymphoma cells (CD19, CD20, etc.) at the different analysis times and/or the median florescence intensity (MFI) of the expression of these markers at the different analysis times and/or the evolution of these percentages and the MFI between 2 analysis times.
  Failure to obtain a complete metabolic response will be defined by: the absence of a complete metabolic response on the PET scans of D30, D90 and M6 in the absence of implementation of a new therapeutic line; or by the absence of complete metabolic response on all PET scans carried out before the implementation of a new therapeutic line.

SECONDARY OUTCOMES:
Identification of a phenotypic "signature" of trogocytosis predictive of the occurrence of grade II or more immunological adverse events | During 60 days after CAR-T cells injection
  Using flow cytometry analysis, the phenotypic "signature" will be assessed by the AUC used to predict the occurrence of immunological side effects (Cytokine Release Syndrome and immune effector cell-associated neurotoxicity syndrome) of grade II or + according to the American Society for Transplantation and Cellular Therapy ASTCT2 criteria. It will be established on circulating CAR-T, T lymphocytes and NK cells of patients, and defined as : the percentage of cells aberrantly expressing different tumor antigens normally expressed on lymphoma cells at the different analysis times,and/or the MFI of the expression of these markers at the different analysis times and/or the evolution of these percentages and the MFI between 2 analysis times.The occurrence of immunological side effects between D0 and D60 will be assessed by clinical and, if necessary, paraclinical examinations (lumbar puncture, brain MRI, etc.). The grade will be evaluated according to the ASTCT2 criteria.
Identification of a phenotypic "signature" of trogocytosis predictive of the occurrence of serious hematological side effects. | Between Day 30 and 6 months after CAR-T cells injection
  Flow cytometry analysis will be performed to determine the level of trogocytosis by effector cells. The phenotypic "signature" of trogocytosis will be assessed by the AUC used to predict the occurrence of serious hematological side effects (grade III or + cytopenias according to Common Terminology Criteria for Adverse Events CTCAE 5.03 between D30 and M6 after injection of anti-CD19 CAR-T cells .It will be established on circulating CAR-T, T lymphocytes and NK cells of patients, and defined as :the percentage of cells aberrantly expressing different tumor antigens normally expressed on lymphoma cells at the different analysis times, and/or the MFI of the expression of these markers at the different analysis times and/or the evolution of these percentages and the MFI between 2 analysis times. The occurrence of hematological side effects between D30 and M6 will be assessed by blood counts. The grade will be evaluated according to the CTCAE v5.03 criteria.
Determination of the trogocytosis level of normal lymphocytes and NK cells in healthy subjects | At enrollment
  Flow cytometry analysis will be performed on each sample on the day of collection (at enrollment), to determine the level of trogocytosis which will be evaluated by simple analysis of the trogocytosis phenotype of normal lymphocytes and NK cells in healthy subjects. This result will be considered as a negative control to determine the phenotypic "signature" of trogocytosis of the primary and secondary outcomes above.

CONTACTS AND LOCATIONS:
Overall Officials: Ludovic GABELLIER, MD, Principal Investigator — Montpellier University Hospital; Florence GALTIER, MD, Principal Investigator — Montpellier University Hospital
Locations (2):
- France (2):
  - Clinical hematology department, University Hospital, Montpellier
  - Clinical Investigation Center, University Hospital, Montpellier